CLINICAL TRIAL: NCT01542229
Title: Improving PTSD Service Delivery for Veterans With Severe Mental Illness
Brief Title: PTSD (PostTraumatic Stress Disorder) Services for Veterans With SMI (Severe Mental Illness)
Acronym: PTSD/SMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 11-306; Pro00013928 (Other: Medical University of South Carolina IRB)
Record Dates: First submitted 2012-02-17; First posted 2012-03-02 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-05

CONDITIONS: Post Traumatic Stress Disorder; Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Major Depression
Keywords: Post Traumatic Stress Disorder; Severe Mental Illness
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Schizophrenia; Psychotic Disorders; Bipolar Disorder; Depressive Disorder, Major; Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: PE + TAU (Experimental): Prolonged Exposure Therapy +Treatment As Usual
  Interventions: Behavioral: Prolonged Exposure for PTSD (PE) + Treatment as Usual (TAU)
- Arm 2: Usual Treatment (Active Comparator): Treatment As Usual
  Interventions: Behavioral: Treatment As Usual (TAU)

INTERVENTIONS:
Behavioral: Prolonged Exposure for PTSD (PE) + Treatment as Usual (TAU) — 12 weekly sessions of Prolonged Exposure in addition to Treatment As Usual
  Arms: Arm 1: PE + TAU
Behavioral: Treatment As Usual (TAU) — Treatment as usual (TAU) will receive support services through the VA potentially inclusive of case management, psychotropic medication management, and/or supportive counseling
  Arms: Arm 2: Usual Treatment

SUMMARY:
As in the general population, there is no clear standard of care within Veterans Affairs Medical Centers for treating posttraumatic stress disorder (PTSD) among individuals with severe mental illness (SMI). This is a considerable issue because trauma, posttraumatic stress disorder (PTSD), and severe psychiatric comorbidity are particularly common among Veterans and this symptom presentation clearly exacerbates the overall course and severity of mental illness. This study is significant in that it proposes to establish the efficacy of a frontline exposure based intervention for posttraumatic stress disorder (PTSD), Prolonged Exposure, for improving critical clinical, quality of life, and cost outcomes among Veterans with severe mental illness (SMI) enrolled in VA healthcare. Collectively, it is anticipated that these data will establish a much needed clinical course of action for what is considered a vulnerable yet highly underserved patient population.

DETAILED DESCRIPTION:
The overarching aim of this proposal is to compare the efficacy of Prolonged Exposure for posttraumatic stress disorder (PTSD) plus treatment as usual (PE+TAU) relative to treatment as usual (TAU) alone using a randomized, between groups, repeated measures design. One hundred fifty six (156) ethnically/racially diverse male and female Veterans with posttraumatic stress disorder (PTSD) and severe mental illness (SMI) will be recruited from the Charleston VA and affiliated Community Based Outpatient Clinics (CBOCs) during the study time frame. For the investigators' study purposes, severe mental illness (SMI) is defined as (1) the presence of a past year Diagnostic Statistical Manual (DSM-IV) Axis I diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or severe depression (2) resulting in persistent impairment in self-care, work, or social functioning. Veterans will be randomized 1:1 to one of two conditions: PE+TAU or TAU. The active intervention phase is 12 weeks. Veterans randomized to treatment as usual (TAU) will receive support services through the VA potentially inclusive of case management, psychotropic medication management, and/or supportive counseling and Veterans randomized to prolonged exposure (PE) plus treatment as usual (TAU) will receive 12 weekly sessions of prolonged exposure (PE) in addition to treatment as usual (TAU). All participants will be assessed at baseline, 6 weeks, post-treatment, and at 3 and 6 months. Additionally, they will complete two self report forms during sessions 3, 6, and 9.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Posttraumatic Stress Disorder (PTSD) on the Clinician Administered PTSD Scale (CAPS; Blake et al., 1990);
* A confirmed diagnosis of a psychotic disorder, bipolar disorder, or severe unipolar depression on the Mini Neuropsychiatric Interview (MINI; Sheehan et al., 1998).

Exclusion Criteria:

* Having a household member who is already enrolled in the study;
* Active psychosis, mania, or dementia at screening;
* Suicidal ideation with clear intent;
* Current substance dependence; and
* Concurrent enrollment in another clinical trial for PTSD or depression.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2012-05-03 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anouk L Grubaugh, PhD MA BS, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grubaugh AL, Tuerk PW, Egede LE, Frueh BC. Perceptions of PTSD research participation among patients with severe mental illness. Psychiatry Res. 2012 Dec 30;200(2-3):1071-3. doi: 10.1016/j.psychres.2012.07.039. Epub 2012 Aug 9. PMID 22884217
- [Result] Brown WJ, Wilkerson AK, Milanak ME, Tuerk PW, Uhde TW, Cortese BM, Grubaugh AL. An examination of sleep quality in veterans with a dual diagnosis of PTSD and severe mental illness. Psychiatry Res. 2017 Jan;247:15-20. doi: 10.1016/j.psychres.2016.07.062. Epub 2016 Sep 30. PMID 27863313
- [Result] Grubaugh AL, Clapp JD, Frueh BC, Tuerk PW, Knapp RG, Egede LE. Open trial of exposure therapy for PTSD among patients with severe and persistent mental illness. Behav Res Ther. 2016 Mar;78:1-12. doi: 10.1016/j.brat.2015.12.006. Epub 2015 Dec 28. PMID 26797658
- See also: pubmed — http://www.ncbi.nlm.nih.gov/pubmed/21596012
- See also: pubmed — http://www.ncbi.nlm.nih.gov/pubmed/28760103
- See also: pubmed — http://www.ncbi.nlm.nih.gov/pubmed/28701969

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: PE + TAU: Prolonged Exposure Therapy +Treatment As Usual
  PE + TAU: 12 weekly sessions of Prolonged Exposure in addition to Treatment As Usual
- Arm 2: Usual Treament: Treatment As Usual
  Treatment As Usual: TAU will receive support services through the VA potentially inclusive of case management, psychotropic medication management, and/or supportive counseling
Period: Overall Study
Arm/Group | Arm 1: PE + TAU | Arm 2: Usual Treament
Started | 68 | 66
Completed | 45 | 30
Not Completed | 23 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: PE + TAU | Arm 2: Usual Treament | Total
Number analyzed (Participants) | 68 | 66 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.33 (12.85) | 46.51 (12.10) | 46.01 (12.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 32
  Male | 50 | 52 | 102

OUTCOME MEASURES:

1. Primary Outcome: Posttraumatic Stress Disorder (PTSD) Checklist (PCL)
Description: The PTSD Checklist (PCL) is a 17-item self-report measure of PTSD symptoms based on DSM-IV criteria. Total scores on the PCL were used, and total scores range from 17 to 85 with higher scores indicative of greater PTSD severity.
Time Frame: pre to post treatment (12 weeks)
Population: Variability in sample size for primary outcomes pre to post due to attrition (i.e., treatment dropout and/or lost to follow-up).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1: PE + TAU | Arm 2: Usual Treament
Number analyzed (Participants) | 35 | 42
score on a scale
  pre treatment (tx) mean | 66.94 (1.71) | 66.33 (1.56)
  post treatment (tx) mean | 51.20 (2.49) | 60.60 (2.27)

2. Primary Outcome: Clinician Administered Posttraumatic Stress Disorder Scale (CAPS)
Description: The Clinician Administered PTSD (Posttraumatic Stress Disorder; PTSD) Scale (CAPS) is a 30-item structured interview that corresponds to DSM-IV criteria for PTSD. The CAPS can be used to make a current (past month) or lifetime diagnosis of PTSD or to assess symptoms over the past week/month. The CAPS was used to measure current PTSD (yes/no diagnosis) as well as total PTSD severity (scores range 0-136, with higher scores indicative of more severe PTSD).
Time Frame: pre to post treatment (12 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Arm 2: Usual Treatment: Treatment As Usual
  Treatment As Usual: TAU will receive support services through the VA potentially inclusive of case management, psychotropic medication management, and/or supportive counseling
Arm/Group | Arm 1: PE + TAU | Arm 2: Usual Treatment
Number analyzed (Participants) | 33 | 45
score on a scale
  pre treatment (tx) mean | 69.00 (2.87) | 62.91 (2.45)
  post treatment (tx) mean | 49.42 (4.42) | 68.42 (3.78)

3. Secondary Outcome: Beck Depression Inventory-II (BDI-II)
Description: The Beck Depression Inventory-II is a 21 item measure of depressive severity. Total BDI-II scores were used. Scores on the BDI-II range from 0 to 63 with higher scores indicative of greater symptom severity.
Time Frame: pre to post treatment (12 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1: PE + TAU | Arm 2: Usual Treatment
Number analyzed (Participants) | 30 | 35
score on a scale
  pre treatmetn (tx) mean | 37.26 (2.08) | 31.54 (1.83)
  post treatment (tx) mean | 26.52 (2.89) | 30.00 (2.53)

4. Secondary Outcome: Brief Psychiatric Rating Scale-Extended (BPRS-E)
Description: The Brief Psychiatric Rating Scale-Extended (BPRS-E) is a 24 item measure of psychopathology across several dimensions (i.e., delusions, motor hyperactivity, withdrawal and blunted affect, self-neglect, etc.) and is a commonly used measure for severely and persistently ill patient populations. Total BPRS scores were used and can range from 24 (score of 1 on all items, symptom not present) to 168 (score of 7 on all items, extremely severe).
Time Frame: pre to post treatment (12 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1: PE + TAU | Arm 2: Usual Treament
Number analyzed (Participants) | 32 | 45
score on a scale
  pre treatment (tx) mean | 47.34 (2.11) | 44.87 (1.78)
  post treatment (tx) mean | 33.72 (1.55) | 35.29 (1.31)

5. Secondary Outcome: Veterans SF 12 Health Survey (SF-12)
Description: The Veterans SF 12 Health Survey (SF-12) is a valid and reliable instrument to measure quality of life and/or functional status in Veterans. The SF-12 was used to track changes in general mental [MCS mental component score) and physical health (PCS physical component score) functioning. Scores on the SF-12 scales range from 0 to 100 once converted and higher scores are indicative of better mental and physical health. The MCS score was used in the current analyses.
Time Frame: pre to post treatment (12 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1: PE + TAU | Arm 2: Usual Treament
Number analyzed (Participants) | 30 | 39
score on a scale
  pre treatment (tx) mean | 36.69 (2.10) | 42.48 (1.78)
  post treatment (tx) mean | 44.31 (2.14) | 42.70 (1.82)

6. Secondary Outcome: Pittsburgh Seep Quality Index
Description: The Pittsburgh Sleep Quality Index (PSQI) is a 19-item commonly used and well validated self-report measure of sleep quality and disturbance. Scores on the PSQI range from 0 to 21, with ratings of 5 or higher indicative of poor sleep quality. Item 9, assessing overall quality of sleep, was used in current analyses. Scores on this item range from 0 to 3, with higher scores indicative of worse sleep quality.
Time Frame: pre to post treatment (12 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1: PE + TAU | Arm 2: Usual Treatment
Number analyzed (Participants) | 32 | 42
score on a scale
  pre treatment (tx) mean | 2.47 (.119) | 2.45 (.103)
  post treatment (tx) mean | 2.00 (.148) | 2.29 (.129)

7. Post Hoc Outcome: Hamilton Depression Scale
Description: The Hamilton Depression Scale (HAM-D) is a 17, 21, or 24 item measure of depression severity. In the 17-item version, which was used, nine of the items are scored on a five-point scale, ranging from 0 to 4; and 8 of the items are scored on a 3-point scale, ranging from 0 to 2. Total scores on the HAM-D are summed and range from 0-53 with higher scores reflective of more severe depressive symptoms.
Time Frame: pre to post treatment (12 weeks)
Population: A subset of participants were administered the HAM-D as an exploratory analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1: PE + TAU | Arm 2: Usual Treatment
Number analyzed (Participants) | 26 | 43
score on a scale
  pre treatment (tx) mean | 18.15 (1.20) | 17.56 (.93)
  post treatment (tx) mean | 10.23 (1.35) | 14.23 (1.05)

8. Post Hoc Outcome: Psychotic Symptom Rating Scales
Description: The Psychotic Symptom Rating Scales (PSYRATS) is an instrument designed to quantify the severity of delusions and hallucinations. The measure has 17 items scored from 0 to 4 (11 items measure auditory hallucinations; 6 items measure delusions). Scores range from 0 to 68 and are summed with higher scores reflective of more severe psychosis.
Time Frame: pre to post treatment (12 weeks)
Population: A subset of participants were administered the HAM-D as an exploratory analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1: PE + TAU | Arm 2: Usual Treatment
Number analyzed (Participants) | 4 | 5
score on a scale
  pre treatment (tx) mean | 30.00 (5.40) | 11.60 (4.83)
  post treatment (tx) mean | 23.00 (8.96) | 16.60 (8.02)

9. Post Hoc Outcome: The Difficulties in Emotion Regulation Scale
Description: The Difficulties in Emotion Regulation Scale (DERS) is a 36-item self-report questionnaire designed to assess multiple aspects of emotion dysregulation. It yields a total score as well as 6 scale scores: Non-acceptance of emotional responses; Difficulties engaging in goal directed behavior; Impulse control difficulties; Lack of emotional awareness; Limited access to emotion regulation strategies; and Lack of emotional clarity. Item scores range from 1 "almost never" to 5 "almost always" with total summed scores ranging from 36 to 180, and higher scores reflective of greater emotion regulation difficulties.
Time Frame: baseline
Population: The DERS was added at a later time as an exploratory variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: PE + TAU | Arm 2: Usual Treatment
Number analyzed (Participants) | 25 | 26
score on a scale | 119.00 (26.08) | 114.15 (26.14)

10. Post Hoc Outcome: Young Mania Scale
Description: The Young Mania Rating Scale (YMRS) is a commonly used measure to assess manic symptoms. The scale has 11 items and is based on the patient's subjective report of his or her clinical condition. Additional information is based upon clinical observations made during the course of the clinical interview. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. Scores range from 0 to 60 and are summed with higher scores reflective of higher symptom severity.
Time Frame: pre to post treatment (12 weeks)
Population: A subset of participants were administered the HAM-D as an exploratory analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1: PE + TAU | Arm 2: Usual Treatment
Number analyzed (Participants) | 15 | 15
units on a scale
  pre treatment (tx) mean | 5.10 (1.54) | 6.91 (1.47)
  post treatment (tx) mean | 3.60 (1.96) | 2.00 (1.86)

ADVERSE EVENTS:
Arm/Group | Arm 1: PE + TAU | Arm 2: Usual Treament
All-Cause Mortality (participants affected / at risk) | 1/68 | 1/66
Serious Adverse Events (participants affected / at risk) | 0/68 | 1/66
Other Adverse Events (participants affected / at risk) | 0/68 | 0/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: PE + TAU (N=68) | Arm 2: Usual Treament (N=66)
psychiatric hospitalization (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes